CLINICAL TRIAL: NCT06219993
Title: Comparison of Robot-assisted Modified Kasai Portoenterostomy With Open Kasai Portoenterostomy for Biliary Atresia
Brief Title: Robot-assisted Modified Kasai Portoenterostomy Versus Open Kasai Portoenterostomy for Biliary Atresia
Acronym: RKPEVSOKPE
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Zunyi Medical College (Other)
Responsible Party: Principal Investigator, zebing Zheng, prof., Zunyi Medical College
Other Study IDs: Robot Kasai Surgery; 82060100 (Other Grant/Funding Number: National Natural Science Foundation of China); ZK-2021-361 (Other Grant/Funding Number: Basic Research Project of Guizhou Province China)
Record Dates: First submitted 2023-12-24; First posted 2024-01-23 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Biliary Atresia; Kasai Operation; Robotic Surgery; Open Surgery
Keywords: biliary atresia; kasai portoenterostomy; Robotic kasai; outcome; RCTs
MeSH Terms: conditions — Biliary Atresia

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RKPE group: 1. Firstly, the Exploring hepatic subcapsular spider-like telangiectasis (HSST) sign at the surface of the liver, and indocyanine green (ICG) cholangiography were observed to confirm the BA diagnosis by Da Vinci robot.
  2. The Roux-en-Y jejunojejunostomy reconstruction was fashioned extracorporeally through the umbilical incision.
  3. With Da Vinci robotic electric scissors help, the fibrous plate was horizontally cut from the middle of the portal plate and transected from to the left and to the right sides which was the Glissonian systems enter the liver parenchyma until see the bile outflow by verified by ICG. The opening of microbile ducts and abundant bile outflow were clearly visible under 10× camera of Da Vinci robot.
  4. Last, an end-to-side hepaticojejunostomy was conducted with one-layer continuous 5-0 PDS sutures posteriorly and anteriorly. A drainage tube was left under the liver, and the incision was closed.
  Interventions: Procedure: robot-assisted modified Kasai portoenterostomy
- OKPE group: 1. The Exploring hepatic subcapsular spider-like telangiectasis (HSST) sign at the surface of the liver, cholangiography were observed to confirm the BA diagnosis by conventional open surgery.
  2. The Roux-en-Y jejunojejunostomy reconstruction by hand-sewn anastomosis.
  3. Dissecting forceps and electric scissors were applied to dissociate the atresia bile ducts and lymph nodes in portal hepatis. Exposed the hepatic artery and portal vein. All portal vein tributaries that drain into the fibrous cone were coagulated by bipolar coagulation to expose the portal plate for resection. With scissors help, the fibrous cone of the hilar region was transected from left to right (the level of transection depends on adequate bile outflow).
  4. Last, an end-to-side hepaticojejunostomy was conducted with one-layer interrupt 5-0 PDS sutures posteriorly and anteriorly. A drainage tube was left under the liver, and the incision was closed.
  Interventions: Procedure: traditional open Kasai portoenterostomy

INTERVENTIONS:
Procedure: robot-assisted modified Kasai portoenterostomy — 1. A 1.0 cm incision was made around the umblilicus for the camera port. 1.Firstly, the Exploring hepatic subcapsular spider-like telangiectasis (HSST) sign at the surface of the liver, and indocyanine green (ICG) cholangiography were observed to confirm the BA diagnosis.
  2. dissecting forceps and electric scissors were applied to dissociate the atresia bile ducts and lymph nodes in portal hepatis. Exposed the hepatic artery and portal vein. All portal vein tributaries that drain into the fibrous cone were coagulated by bipolar coagulation to expose the portal plate for resection. With electric scissors help, the fibrous plate was horizontally cut from the middle of the portal plate and transected from to the left and to the right sides which was the Glissonian systems enter the liver parenchyma until see the bile outflow by verified by ICG. The opening of microbile ducts and abundant bile outflow were clearly visible under 10× camera of Da Vinci robot.
  Groups: RKPE group
Procedure: traditional open Kasai portoenterostomy — Dissecting forceps and electric scissors were applied to dissociate the atresia bile ducts and lymph nodes in portal hepatis. Exposed the hepatic artery and portal vein. All portal vein tributaries that drain into the fibrous cone were coagulated by bipolar coagulation to expose the portal plate for resection. With scissors help, the fibrous cone of the hilar region was transected from left to right (the level of transection depends on adequate bile outflow).
  Groups: OKPE group

SUMMARY:
Open Kasai portoenterostomy (OKPE) is considered the standard treatment procedure for biliary atresia (BA). Robotic-assisted Kasai portoenterostomy (RAKPE) has been utilized to treat BA. However, there were no randomized controlled trials to verify its effectiveness. The objection was to compare the efficacy of Da Vinci robot-assisted with open Kasai portoenterostomy for biliary atresia.

DETAILED DESCRIPTION:
Biliary atresia (BA) is one of the most common cholestatic childhood diseases, with an estimated incidence of 1 in 8000-18,000 live births. BA is a progressive cholangiopathy with fibro-obliterative obstruction of the bile duct. The exact pathogenesis and etiology of BA have not been fully elucidated. The hypothesis that is most widely recognized states that injury to the biliary duct is caused by an initial infection and then an autoimmune response is induced by infection, leading to progressive damage to the biliary duct. Typical clinical manifestations of BA include persistent jaundice, acholic stools, and pigmented urine in the first months after birth. Unfortunately, the presentation time of the clinical features can be delayed in BA, which may lead to misdiagnosis. The average diagnostic age of BA is 60 days in many countries. Currently, effective management for BA is the Kasai portoenterostomy (KPE), which was originally reported by Morio Kasai in 1959. open Kasai portoenterostomy (OKPE) has been introduced to restore bile drainage for patients with BA and become the gold standard. Esteves et al. reported laparoscopic Kasai portoenterostomy (LKPE) for BA in 2002, but its efficacy remains controversial compared with OKPE. Several centers have revealed positive results with modified LKPE procedures. Nonetheless, LKPE is still a complex and challenging procedure with difficulties in fiber block dissection and anastomosis, resulting in a long learning curve. With merits of articulating wrists, 3D imaging field of vision and filter tremor, robotic surgery has been gradually applied to hepatobiliary disorders in children. Theoretically, robotic-assisted Kasai portoenterostomy (RAKPE) may overcome the difficulties of LKPE in fiber block dissection and anastomosis, thereby becoming a better option for BA. Currently, reports of RAKPE in infants with BA are limited to small case series, and its effectiveness remains controversial. However, there were no randomized controlled trials to verify its effectiveness. The objection was to compare the efficacy of Da Vinci robot-assisted with open Kasai portoenterostomy for biliary atresia.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosis type Ⅲ biliary atresia who underwent open kasai portoenterostomy or robotic-assisted Kasai portoenterostomy, aged no more than 6 months.

Exclusion Criteria:

* TypeⅠbiliary atresia and typeⅡbiliary atresia. biliary atresia combined with severe cardiopulmonary diseases.

Max Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: patients diagnosis type Ⅲ biliary atresia who underwent open kasai portoenterostomy or robotic-assisted Kasai portoenterostomy, aged no more than 6 months.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-12-21 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Survival native liver rate(%) | 2 years
  1- and 2-year survival with native liver (SNL) were recorded.
Jaundice clearance rate(%) | 6 months, 1 year and 2 years
  Jaundice clearance (JC) was defined as serum total bilirubin level ≤ 20 μmol/L (or ≤ 1.2 mg/dL) within 6 months after the Kasai operation. JC within 6 months after surgery is widely used as the accepted measure of successful Kasai portoenterostomy.

SECONDARY OUTCOMES:
Incidence of Cholangitis (%) | 2 years
  Cholangitis was defined as having more than two clinical presentations [fever (> 38 °C) or stool color change or increased/increasing jaundice] and two laboratory tests [elevated inflammatory parameters or increased/increasing transaminases or increased/increasing gamma-glutamyl transferase (GGT)/ bilirubin].
Operative time (min) | 1 year
  The operative time(minute) in two groups
Estimated blood loss(ml) | 1 year
  The surgeon estimated blood loss(ml) in two groups
Bile leakage rate (%) | 1 year
  The incidence of complication of bile leakage between two groups.
Time to enteral feeding (days) | 1 year
  The time patients from operation to the first oral feeding
Postoperative hospital stay (days) | 6 months
  we record the times of postoperative hospital stay
Wound infection (%) | 1 year
  The incidence of complication of wound infection between two groups
Variceal bleeding rate(%) | 2 years
  The incidence of complication of Variceal bleeding between two groups.
Volvulus (%) | 1 year
  the incidence of Volvulus with adhesive bands and malrotation because of anastomotic ileus in two groups after operation 1year
Time to drain removal (days) | 6 months
  we record the time of drain removal
Umbilical hernia rate（%） | 1 year
  The incidence of complication of umbilical herniabetween two groups
Blood transfusion in theperioperative period (ml) | 6 months
  the blood transfusion in theperioperative period
C-reactive protein level (mg/dl) | 6 months
  C-reactive protein level at POD 1

OTHER OUTCOMES:
Jaundice-free survival with a native liver rate (%) | 2 years
  Jaundice-free survival with a native liver in 6 months,1 year and 2 years
Survival with liver transplantation rate (%) | 2 years
  Survival with liver transplantation in 6 months, 1year and 2 years.
Died (%) | 2 years
  we record the incidence of died at 6 months, 1year and 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhu Jin, MD, Study Chair — Zunyi Medical College
Locations (2):
- China (2):
  - Affiliated Hospital of Zunyi Medical University, Zunyi, Guizhou
  - Affiliated hospital of zunyi medical university, Zunyi, Guizhou

IPD SHARING:
Plan to Share IPD: No
The individual participant in this study we recruit are mainly minors, which involves privacy protection for minors, so we cannot share the personal information of participants to the other researchers.

REFERENCES:
- [Result] Zhang M, Cao G, Li X, Zhang X, Li Y, Chi S, Rong L, Tang ST. Robotic-assisted Kasai portoenterostomy for biliary atresia. Surg Endosc. 2023 May;37(5):3540-3547. doi: 10.1007/s00464-022-09855-x. Epub 2023 Jan 5. PMID 36602550
- [Result] Murase N, Hinoki A, Shirota C, Tomita H, Shimojima N, Sasaki H, Nio M, Tahara K, Kanamori Y, Shinkai M, Yamamoto H, Sugawara Y, Hibi T, Ishimaru T, Kawashima H, Koga H, Yamataka A, Uchida H. Multicenter, retrospective, comparative study of laparoscopic and open Kasai portoenterostomy in children with biliary atresia from Japanese high-volume centers. J Hepatobiliary Pancreat Sci. 2019 Jan;26(1):43-50. doi: 10.1002/jhbp.594. Epub 2019 Jan 12. PMID 30488647